CLINICAL TRIAL: NCT06958926
Title: A Translational Study for Locoregional Recurrence of T4 Colon Cancer
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202407175RINC
Record Dates: First submitted 2025-04-14; First posted 2025-05-06 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: T4 Colorectal Cancer; Colorectal Cancer Stage III; Colorectal Cancer Stage II
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ascites cell-free DNA, serum cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radical surgery for colon and rectum cancer — Radical surgery for colon and rectum cancer indicates that the surgery intends to eradicate all identifiable tumor in the human body.
Procedure: Radical surgery for colorectal cancer — Radical surgery for colorectal cancer indicates that the surgery intends to eradicate all identifiable tumor in the human body.

SUMMARY:
The outcome of T4 locally advanced colon cancer is poor when locoregional recurrence occurred. Previous studies had showed that the aggravation of T4 colon cancer is higher than N-positive colon cancer, contributing to staging paradox that outcomes of stage IIB/C are poorer than stage IIIA colon cancer and higher locoregional recurrence of stage IIB/C colon cancer. The phenomenon cannot be explained by radicality, lymph node harvested and adjuvant chemotherapy administration. To elucidate the cancerous aggravation of T4 colon cancer, the investigators should dive into the clinicopathology, metastatic mechanism and cancer biology.

The investigators hypothesize that peritoneal spreading can be one of the metastatic routes of T4 colon cancer; however, few studies have addressed the finding and deserved investigation. Previous research have found that serum epigenetic alterations and cell-free DNA can serve as a prognostic marker for stage II/III colon cancer.

Therefore, the aim of this study is (1) to explore the role of ascites cfDNA as a potential biomolecular marker for locoregional recurrence; (2) to identify the risk factors of locoregional recurrence for T4 colon cancer by correlating biomolecular markers between clinicopathology, epigenomic alterations in blood and ascites.

ELIGIBILITY:
* Inclusion Criteria:

  1. Age ≥ 18 years old
  2. Diagnosed as colorectal cancer
  3. Undergo radical colectomy or palliative colectomy, not limited to minimally invasive surgery or open surgery
* Exclusion Criteria:

  1. Age<18 years old
  2. Pregnancy
  3. Patients with peritoneal dialysis
  4. Patients who are unwilling to undergo colorectal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected cT4 or pT4 colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The correlation the cell-free DNA level and sequencing between ascites and serum | One year

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Tso Liao, MD, PhD, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch; Yu-Tso Liao, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided